CLINICAL TRIAL: NCT05943912
Title: Myopia Control Effect of DIMS Spectacle Lenses in Czech Children and Young Adults
Status: Active, not recruiting | Type: Observational
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Other Study IDs: SGS23/195/OHK4/3T/17
Record Dates: First submitted 2023-07-04; First posted 2023-07-13 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Myopia
Keywords: myopia; axial length; DIMS
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single Vision Spectacle Lens: Participants who chose to correct myopia with single vision spectacle lenses.
  Interventions: Other: Single Vision Spectacle Lens
- Defocus Incorporated Multiple Segments (DIMS) Spectacle Lens: Participants who chose to correct myopia with DIMS spectacle lenses.
  Interventions: Other: Defocus Incorporated Multiple Segments (DIMS) Spectacle Lens

INTERVENTIONS:
Other: Single Vision Spectacle Lens — 36 months of therapy
  Groups: Single Vision Spectacle Lens
Other: Defocus Incorporated Multiple Segments (DIMS) Spectacle Lens — 36 months of therapy
  Groups: Defocus Incorporated Multiple Segments (DIMS) Spectacle Lens

SUMMARY:
The aim of this clinical study is to compare the efficacy of DIMS technology spectacle lenses with conventional single vision spectacle lenses at slowing the progression of myopia in the category of children and young adults during three years.

DETAILED DESCRIPTION:
The study is non randomized, unmasked, observational and prospective. Participants aged 6-26 with progressing myopia (but no ocular pathology), all Caucasian, are divided in two groups according to single vision spectacle lenses (SV) and DIMS technology lenses (DIMS). The participants are followed during three years (axial length, refraction changes).

Defocus incorporated multiple segments (DIMS) spectacle lenses were designed to slow myopia progression in children, based on the principle of peripheral myopic defocus. DIMS spectacles reduce the progression of myopia and reduce axial elongation by 50-60% compared to single vision (SV) lenses according to previous scientific studies conducted mostly on the Asian population under the age of 15.

The majority of myopia appears and progresses during childhood. The myopia stabilizes by the age of 18 years, a number of individuals may still present myopic changes.

The goals of our study:

* compare the efficacy of DIMS spectacle lenses with SV spectacle lenses at slowing the progression of myopia in the category of Czech children and young adults (effect on axial length and refractive changes)
* monitoring axial length and refractive changes in myopic children and young adults (aged 6-26)
* monitoring adaptation to DIMS lenses in myopes aged 6-26 years monitoring the influence of the environment and individual behavior on the progression of myopia

ELIGIBILITY:
Inclusion Criteria:

* Progressive myopia
* Myopes aged 6-26 years
* Myopia between -0,25D and -8,5D
* Astigmatism -0,25 and -2,25DC

Exclusion Criteria:

* Ocular pathology
* Amblyopia
* Strabism
* Non-compliance to eye examinations

Ages: 6 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: To evaluate the efficacy of Defocus Incorporated Multiple Segment (DIMS) lenses in slowing myopia progression in a young European population of progressing myopes. A prospective, non-randomized, observational 3 - year study will be conducted in 80 progressing myopes aged 6-26 years, with myopia between -0,25D and -8,5D and astigmatism -0,25 and -2,25DC. Participants self-selected wearing DIMS (n=55) or single vision (SV) lenses (n=25). Spherical Equivalent Refraction (SER, cycloplegic autorefraction) and axial length (AL) were measured at baseline. AL will be measured at 3M, 6M and every 6M and SER will be measured every 12M.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Axial length of eye | in 36 moths therapy
  biometry (Lenstar 900)

SECONDARY OUTCOMES:
Objective refraction | in 36 month therapy
  autorefractometer (Huwitz)

CONTACTS AND LOCATIONS:
Overall Officials: Marketa Zakova, Ph.D., Study Director — Czech Technical University in Prague
Locations (1):
- Czech Technical University, Prague, Czech Republic, Czechia